CLINICAL TRIAL: NCT03678259
Title: Evaluation of 124I-p5+14 Injection as an Imaging Agent for the Detection of Systemic Amyloidosis
Brief Title: 124I-p5+14 Injection Safety in Subjects With Systemic Amyloidosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AMY1001
Record Dates: First submitted 2018-07-30; First posted 2018-09-19 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2021-07

CONDITIONS: Systemic Amyloidosis
Keywords: Amyloidosis, AL, ATTR, ALect2
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis

STUDY DESIGN:
Intervention Model Description: The first three patients enrolled in the trial (Part 1) will take part in a dose-escalation study and will receive a single IV dose 11.1 MBq (0.3 mCi; n = 1), 37 MBq (1 mCi; n = 1) or 74 MBq (2 mCi; n = 1) of 124I-p5+14 Injection. The trial then will be opened to include another 54 patients who will receive a single IV bolus injection of 2 mCi 124I-p5+14 Injection. Every patient participating will receive < 2 mg of peptide p5+14. The study comprises five parts.In Part 2, the trial will enroll SA patients with confirmed AL, ATTR, ALECT2, or other forms of amyloidosis.In Part 3, the trial will study asymptomatic subjects with genetically confirmed mutation of the transthyretin gene.Part 4 will include five healthy control subjects.Part 5 will recruit previously enrolled subjects from Parts 2 or 3 who received a 2 mC dose of 124I-p5+14 Injection and had images confirming the presence of abnormal amyloid deposits for a second exposure to 124I p5+14 Injection and second PET/CT scan.
Masking Description: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 124I-p5+14 Injection (Experimental): A single-injection dose of 124I-p5+14 adequate for imaging amyloid deposits by using PET/CT imaging in subjects with confirmed systemic amyloidosis of several sub-types.
  Interventions: Drug: 124I-p5+14 Injection

INTERVENTIONS:
Drug: 124I-p5+14 Injection — 124I-p5+14 Injection which is a formulation of a synthetic, all natural, 45 amino acid peptide (MW = 4766.4) with a net +12 positive charge
  Other Names: APi1832

SUMMARY:
This is a single-center, exploratory, Phase 1 Positron Emission Tomography/x-ray Computed Tomography (PET/CT) imaging study to detect amyloidosis that will enroll patients with a confirmed diagnosis of systemic amyloidosis. The purpose of this exploratory trial is to assess the safety and efficacy of 124I-p5+14 Injection at a single-injection dose adequate for imaging amyloid deposits by using PET/CT imaging in subjects with confirmed systemic Immunoglobulin Light Chain-associated Amyloidosis (AL), Transthyretin-associated Amyloidosis (ATTR), Leukocyte Chemotactic Factor 2-associated Amyloidosis (ALect2) as well as other types.

DETAILED DESCRIPTION:
The rationale for this study is the discovery of a synthetic polypeptide, designated p5+14, a synthetic 45 amino acid peptide that binds many forms of amyloid, including human AL-, ATTR- and ALect2-associated amyloid, as well as human and murine serum amyloid protein A-associated (AA) amyloid. In preclinical studies, using SPECT and PET imaging, as well as microautoradiography, it has been shown that radioiodinated p5+14 binds rapidly and specifically to all amyloid deposits in abdominothoracic organs and tissues.

This is a single site, exploratory, open-label Phase I PET/CT imaging and dosimetry study. The investigational drug product (designated 124I-p5+14 Injection) is an amyloid-reactive synthetic peptide, p5+14 (also known as APi1832), radiolabeled with iodine-124 (I-124 or 124I). All patients enrolled in this exploratory trial will be outpatients with a confirmed diagnosis of systemic amyloidosis.

The first three patients enrolled in the trial (Part 1) will take part in a dose-escalation dosimetry study and will receive a single intravenous (IV) dose of 11.1 Megabecquerel (MBq) (0.3 millicuries (mCi); n = 1), 37 MBq (1 mCi; n = 1) or 74 MBq (2 mCi; n = 1) of 124I-p5+14 Injection for the purpose of determining estimates of organ-associated and whole body radioactive dosimetry.

The trial then will be opened to include another 54 patients who will receive a single IV bolus injection of 2 mCi 124I-p5+14 Injection. Every patient participating will receive < 2 mg of peptide p5+14. The study comprises five parts.

In Part 2, the trial will enroll SA patients with confirmed AL, ATTR, ALECT2, or other forms of amyloidosis.

In Part 3, the trial will study asymptomatic subjects with genetically confirmed mutation of the transthyretin gene.

Part 4 will include five healthy control subjects. Part 5 will recruit previously enrolled subjects from Parts 2 or 3 who received a 2 mC dose of 124I-p5+14 Injection and had images confirming the presence of abnormal amyloid deposits for a second exposure to 124I p5+14 Injection and second PET/CT scan.

ELIGIBILITY:
Subjects included in this trial are volunteers with a confirmed diagnosis of systemic amyloidosis, a genetically well-defined mutation of the TTR gene but without clinical evidence of active disease, and at an age typical of development of symptomology ≥ 50, or healthy control subjects (≥30 years).

Prior to participation in Parts 1 or 2 of the trial (n = 73), the following inclusion criteria must be met

Subjects included in this trial are volunteers with a confirmed diagnosis of systemic amyloidosis, a genetically well-defined mutation of the TTR gene but without clinical evidence of active disease, and at an age typical of development of symptomology ≥ 50, or healthy control subjects (≥30 years).

Prior to participation in Parts 1 or 2 of the trial (n = 73), the following inclusion criteria must be met:

1. Patients must have a confirmed diagnosis of systemic amyloidosis, based on either a histologic confirmation that a biopsy contains deposits of apple-green birefringent, Congophilic material or genetic screening and presence of amyloid-related pathology, or amyloid-specific imaging study. Additionally, the type of amyloidosis (AL, ATTR, ALect2, or other) should be characterized.
2. Patients enrolled in Part 1 (n = 3) must have widespread AL amyloidosis, defined as biopsy proven or clinically detectable involvement, of at least two organs (excluding the peripheral nervous system).
3. All patients in Parts 1 and 2 will be 18 years of age or older. There are no gender or racial restrictions.
4. Women of child bearing potential (those who have not been surgically sterilized, are not postmenopausal [typically understood to mean last menstrual period >2 y ago without pharmaceutical intervention], and women who are fertile) must test negative for pregnancy in a laboratory test administered by the site physician.
5. Patients who have had or are currently receiving therapy or other drug based anti-amyloid regimens can be included on study (Parts 1 and 2).
6. Patients must provide signed, written, informed consent and be willing to comply with eligibility requirements, scheduled visits, and follow-up studies.
7. Due to annual dosimetry limitations, patients who have participated in another nuclear medicine amyloid imaging clinical trial protocol can be included in this study no earlier than 12 months after the previous radiotracer injection.
8. In Part 2, inclusion of patients with amyloid subsets AL, ATTR, and ALect2 will continue until the trial has achieved recruitment goals for each subset: 30 AL; 20 ATTR; 5 ALect2; and 10 15 "Other".

Prior to participation in Part 3 (n = 10 subjects) of the trial, the following inclusion criteria must be met:

1. Patients must have a well-defined germline mutation of the transthyretin (TTR) gene rendering them at risk for amyloidosis, and be free of clinical evidence of SA.
2. All patients in Part 3 will be >50 years of age. There are no gender or racial restrictions.
3. Women of child bearing potential (those who have not been surgically sterilized, are not postmenopausal [typically understood to mean last menstrual period >2 y ago without pharmaceutical intervention], and women who are fertile) must test negative for pregnancy in a laboratory test administered by the site physician.
4. Subjects must provide signed, written, informed consent and be willing to comply with eligibility requirements, scheduled visits, and follow-up studies.
5. Due to annual dosimetry limitations, subjects who have participated in another nuclear medicine amyloid imaging clinical trial protocol can be included in this study no earlier than 12 months after the previous radiotracer injection.

Prior to participation Part 4 of the trial (n = 5), the following inclusion criteria must be met:

1. Healthy Control Subjects (HC) will be generally healthy adults, either male or female, and will not have a diagnosis of amyloidosis, will not have a first- or second-degree relative (parent, sibling, child, aunt, uncle, niece, nephew) with confirmed or suspected familial amyloidosis, and will not have diabetes mellitus (type 2).
2. All Part 4 subjects will be > 30 years of age or older.
3. Women of child bearing potential (those who have not been surgically sterilized, are not postmenopausal [typically understood to mean last menstrual period >2 y ago without pharmaceutical intervention], and women who are fertile) must test negative for pregnancy in a laboratory test administered by the site physician.
4. Patients must provide signed, written, informed consent and be willing to comply with eligibility requirements, scheduled visits, and follow-up studies.
5. Due to annual dosimetry limitations, patients who have participated in another nuclear medicine imaging clinical trial protocol can be included in this study no earlier than 12 months after the previous radiotracer injection.

Prior to participation in Part 5 of the trial, the following inclusion criteria must be met:

1. Patients must have successfully completed participation in Part 2 or Part 3 of this trial with CT/PET images confirming the presence of abnormal amyloid deposits in thoracoabdominal organs.
2. Patients must have received a 2 mCi dose of 124I-p5+14 Injection during Part 2 or 3 of this trial with visual evidence of uptake of radiotracer in abdominothoracic organs associated with amyloid.
3. The repeat exposure to the study agent must occur at least 6 months after the first exposure.
4. Patients must submit a serum specimen for exploratory evaluation of the presence of anti-p5+14 peptide antibodies, with results reviewed by the Principal Investigator prior to a second exposure to the study agent.
5. The patient must meet all of the Inclusion criteria for participation in Part 2 or Part 3 outlined in Sections 5.2 or Section 5.3 (as applicable), including the signing of an informed consent for Part 5.

In addition, the following criteria will exclude candidates from participation in the trial, Parts 1 and 2:

1. Those with significant co-morbidity (e.g., Eastern Cooperative Oncology Group [ECOG] score of 3 or greater), uncontrolled infection, or other serious illness.
2. Patients with a sustained SpO2 of ≤ 92% as noted in the medical record.
3. Patients that require renal dialysis.
4. Women who are of child bearing potential (those who have not been surgically sterilized, are not postmenopausal [typically understood to mean last menstrual period >2 y ago without pharmaceutical intervention], and women who are fertile) who test positive for pregnancy in a laboratory test administered by the site physician, are pregnant, or are nursing
5. Patients who have received any amyloidophilic radiotracer as part of a research clinical trial (not standard of care) within the past 12 months.
6. Patients with exposure to heparin, or heparin-based medications, within 7 days prior to the imaging study.
7. Patients who have a known allergy to acetaminophen or iOSAT iodine treatment.

The following criteria will exclude candidates from participation in Part 3 of the trial:

1. Those with significant co-morbidity (e.g., Eastern Cooperative Oncology Group [ECOG] score of 3 or greater), uncontrolled infection, or other serious illness.
2. Subjects with a sustained SpO2 of ≤ 92% as noted in the medical record.
3. Women who are of child bearing potential (those who have not been surgically sterilized, are not postmenopausal [typically understood to mean last menstrual period >2 y ago without pharmaceutical intervention], and women who are fertile) who test positive for pregnancy in a laboratory test administered by the site physician, are pregnant, or are nursing.
4. Subjects who have clinical evidence of amyloidosis based on standard clinical criteria.
5. Subjects with polyneuropathy of unknown origin.
6. Subjects who have received any amyloidophilic radiotracer as part of a research clinical trial (not standard of care) within the past 12 months.
7. Subjects with exposure to heparin, or heparin-based medications, within 7 days prior to the imaging study.
8. Subjects who have a known allergy to acetaminophen or iOSAT iodine treatment.
9. Subjects with clinical signs of SA based on routine investigation of serum and urine biomarkers, radiographic or nuclear imaging studies, or peripheral nerve evaluations.

The following criteria will exclude subjects from participation in Part 4:

1. Those with significant co-morbidity (e.g., Eastern Cooperative Oncology Group [ECOG] score of 2 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light house work, office work) or greater), uncontrolled infection, or other serious illness.
2. Individuals with a sustained SpO2 of ≤ 92% as noted in the medical record.
3. Women who are of child bearing potential (those who have not been surgically sterilized, are not postmenopausal [typically understood to mean last menstrual period >2 y ago without pharmaceutical intervention], and women who are fertile) who test positive for pregnancy in a laboratory test administered by the site physician, are pregnant, or are nursing.
4. Subjects who have received any amyloidophilic radiotracer as part of a research clinical trial (not standard of care) within the past 12 months.
5. Subjects with exposure to heparin, or heparin-based medications, within 30 days prior to the imaging study.
6. Subjects who have a known allergy to acetaminophen or iOSAT iodine treatment.
7. Subjects with a diagnosis of Type 2 diabetes mellitus or who are taking medication for management of Type 2 diabetes mellitus.
8. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1.
9. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis.
10. Uncontrolled hypertension (BP > 160/100 mm Hg).
11. Smokes >20 cigarettes a day.
12. A diagnosis of heart failure with preserved ejection fraction.
13. Has any other conditions, which, in the opinion of the Investigator would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the study

The following criteria will exclude subjects from participation in Part 5.

1. Any patient who experienced a clinically significant adverse event related to prior exposure to the study agent.
2. Any subject who meets any of the Exclusion Criteria for Part 2 or Part 3 (as applicable), described in Section 5.3.1 and Section 5.3.2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Organ-specific radioactivity dosimetry (Part 1). | Through 48 hours
  Localization of 124I-p5+14 will be taken from PET/CT images performed at intervals during the 48 hours after injection. Organ-specific dosimetry and whole body dose measurements will be made using Olinda software (Olinda/Exp; Organ Level Internal Dose Assessment/Exponential Modeling)

SECONDARY OUTCOMES:
Absolute values and changes from baseline in clinical laboratory values. | Baseline and 24 hours
  Laboratory assessments will include hematology and clinical chemistry.
Clinically defined amyloidosis organ involvement. | Baseline
  For each subject, the clinician/investigator will designate each organ as involved or not involved with amyloidosis, based on available medical history including prior imaging, prior biopsy results, and clinical laboratory values.
Measure of background radioactivity uptake. | 6 hours and 24 hours
  For each subject, a background radioactivity uptake measure will be derived from the PET images at an uninvolved anatomic site (the lumen of a large blood vessel).
Measure of radioactivity uptake by each organ | 6 hours and 24 hours
  Uptake of 124I-p5+14 will be derived from PET/CT scans performed at 6 hours and 24 hours after injection. Any organ with >=2-fold higher accumulation of radiotracer, relative to the background uptake, will be considered positive.
Concentration of radiotracer in specific anatomic sites, for each subject and anatomic site | 6 hours and 24 hours
  Concentration of 124I-p5+14 will be derived from PET/CT scans performed at 6 hours and 24 hours after injection.
Organ and tissue-specific sensitivity of the 124I-p5+14 Injection radiotracer | 6 hours and 24 hours
  Sensitivity for each organ will be derived from the list of clinically involved organs (Secondary Measure 1) and the list of organ radioactivity uptake (Secondary Measure 4), using the formula, true positive rate = [True positive/(True positive + False negative)].
Correlation between concentration of the radiotracer (Bq/cc) in the kidney with organ-associated clinical biomarkers. | 6 hours and 24 hours
  Statistical correlation of kidney radiotracer uptake with proteinuria, albuminuria, creatinine, and blood urea nitrogen (BUN).
Correlation between concentration of the radiotracer (Bq/cc) in the heart with organ-associated clinical biomarkers. | 6 hours and 24 hours
  Statistical correlation of heart radiotracer uptake with N-terminal-pro-brain natriuretic peptide (NT-BNP) or Brain Natriuretic Peptide (BNP) serum levels, intraventricular septal thickness, and ejection fraction (measures as available from medical history)
Peptide uptake in the heart. | 6 hours and 24 hours
  Peptide uptake will be recorded as the Standard Uptake Value (SUV) or as Bq/cc of organ volume; obtained from the Region of Interest (ROI) analysis
Peptide uptake in the kidney | 6 hours and 24 hours
  Peptide uptake will be recorded as the Standard Uptake Value (SUV) or as Bq/cc of organ volume; obtained from the Region of Interest (ROI) analysis.
Peptide uptake in organ(s) other than kidney or heart if clinically relevant | 6 hours and 24 hours
  Peptide uptake will be recorded as the Standard Uptake Value (SUV) or as Bq/cc of organ volume; obtained from the Region of Interest (ROI) analysis
Correlation between uptake of peptide and clinical status of kidney, heart and other organs | Baseline and 24 hours
  Correlation between uptake of peptide (from ROI measurements) and the clinical status of kidney, heart, and other organs if indicated (clinical status defined as in Secondary Endpoint 1).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Wall, Ph.D., Principal Investigator — UTHSC Graduate School of Medicine
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wall JS, Martin EB, Endsley A, Stuckey AC, Williams AD, Powell D, Whittle B, Hall S, Lambeth TR, Julian RR, Stabin M, Lands RH, Kennel SJ. First in Human Evaluation and Dosimetry Calculations for Peptide 124I-p5+14-a Novel Radiotracer for the Detection of Systemic Amyloidosis Using PET/CT Imaging. Mol Imaging Biol. 2022 Jun;24(3):479-488. doi: 10.1007/s11307-021-01681-2. Epub 2021 Nov 16. PMID 34786667